CLINICAL TRIAL: NCT06693557
Title: Feeding Intolerance in Preterm Infant ,Rate of Occurrences, Risk Factors , Outcomes
Brief Title: Feeding Intolerance in Preterm Infant
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hager Amer Nadi Abdelaziz, 71515,Assiut, Assiut University
Other Study IDs: Feeding intolernce
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Feeding Intolernce

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To determine the incidence and risk factors of feeding intolerance in preterm infants. To assess the outcome of feeding intolerance in preterm infants.

DETAILED DESCRIPTION:
Premature infants frequently suffer from feeding intolerance related to prematurity and are highly associated with morbidity and mortality. [1] Feeding intolerance (FI) is defined as difficulty to digest enteral feedings and is accompanied by an increase in gastric residuals, abdominal distension, and/or reflux. It is common in preterm infants and commonly results in feeding and gastrointestinal disruptions. FI in newborns can be a sign of a variety of problems, ranging from minor, self-limiting illnesses to serious, life-threatening illnesses. [2] The common cause of FI is low intestinal motility because of prematurity , Enzymatic digestion, bacterial colonization, hormonal response, and local immunity are also possible reasons for FI. [3] FI is very common among preterm infants and its clinical symptoms include abdominal distension, vomiting, bilious gastric residuals, occult or gross bloody stools, and are observed in nearly 29% of such neonates. [4] Factors that contribute to feeding intolerance include poor coordination of sucking and swallowing, incompetent lower esophageal sphincter, small gastric capacity, delayed gastric emptying time, and intestinal hypomotility. Abnormal bacterial colonization may be a coexisting factor in feeding intolerance in newborns mainly due to dysfunction of the intestinal barrier, the immune responses, and sensory motor functions of the gut. [5] Mother's milk feeding is related to better feeding tolerance and may be correlated to a reduction in severe morbidity. [6] The mode of delivery (vaginal or cesarean section) and feeding type (breastfeeding or formula feeding) of neonates are considered the most influential factors in the development of gut microbiota. [7] In the preterm infant, the readiness to tolerate enteral nutrition relies upon the degree of maturation of gastro-intestinal (G-I) functions (motility, enzymatic digestion, hormonal responses, bacterial colonization and local immunity). Anatomical development of the GI tract is largely completed at 20 weeks of gestation, although the elongation of the GI tube and increases in the absorbing area (microvilli) continue during the last trimester of gestation and beyond. [8] Successful establishment of enteral feedings is a major goal in the treatment of very low-birthweight infants, but functional immaturity of the gastrointestinal tract may hamper such efforts. Prokinetic agents often are used in an attempt to overcome functional immaturity by speeding up gastric empyting and increase intestinal wall motility.[9]

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants (gestational age < 37 weeks).
* Preterm infants from day 0 to day 28 of life.

Exclusion Criteria:

* We will exclude those babies:
* Full-term babies (gestational age > 37 weeks).
* Preterm babies with gastrointestinal anomalies.
* Preterm babies with suspected inborn errors of metabolism.
* Preterm babies with suspected necrotizing enterocolitis and sepsis at the onset of feeding.

Ages: 1 Week to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants less than 37 weeks
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence and risk factors of feeding intolerance in preterm infants. To assess the outcome of feeding intolerance in preterm infants | Baseline
  To determine the incidence and risk factors of feeding intolerance in preterm infants.by assessment of extremely low birth with congenital heart disease by echo , Respiratory distress syndrome by chest x ray In order to determine : A_ Daily weight gain by BMI B_ Days to reach fulfill feeding C_ Duration of hospital stay.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ford SL, Lohmann P, Preidis GA, Gordon PS, O'Donnell A, Hagan J, Venkatachalam A, Balderas M, Luna RA, Hair AB. Improved feeding tolerance and growth are linked to increased gut microbial community diversity in very-low-birth-weight infants fed mother's own milk compared with donor breast milk. Am J Clin Nutr. 2019 Apr 1;109(4):1088-1097. doi: 10.1093/ajcn/nqz006. PMID 30982856